CLINICAL TRIAL: NCT05026775
Title: Effectiveness and Cost-effectiveness of the Initial Medication Adherence Intervention: Cluster-randomized Controlled Trial and Economic Model
Brief Title: Effectiveness and Cost-effectiveness of the Initial Medication Adherence Intervention
Acronym: IMA-cRCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundació Sant Joan de Déu (Other)
Collaborators: Institut Català de la Salut (Other); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Parc Sanitari Sant Joan de Déu (Other); CIBER of Epidemiology and Public Health (Unknown); Consell de Col·legis de Farmacèutics de Catalunya (Unknown); Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC) (Other)
Responsible Party: Principal Investigator, Maria Rubio-Valera, Head of Quality and Patient Safety, Parc Sanitari Sant Joan de Déu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 948973
Record Dates: First submitted 2021-07-23; First posted 2021-08-30 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Adherence, Medication
Keywords: Complex Intervention; Real World Data; Cardiovascular Disease; Diabetes Mellitus
MeSH Terms: conditions — Medication Adherence; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participant: The randomization is conducted at the primary care centre level. Patients from intervention areas will receive enhanced care but will not be aware of the group assigned.
  Investigator: Data analysists will not have information on which group is the intervention group when conducting the analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Initial Medication Adherence (IMA) intervention (Experimental): General practitioners (GP) will apply the IMA intervention to all patients receiving a new prescription for treatment of cardiovascular disease or diabetes. Following the IMA intervention, nurses and community pharmacists will offer information support in line with the information provided by the GP.
  Interventions: Behavioral: Initial Medication Adherence (IMA)
- Usual care (Active Comparator): Patients will receive the usual care when being prescribed a new prescription for treatment of cardiovascular disease or diabetes. Nurses and community pharmacists will be asked to also provide usual care to those patients.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Initial Medication Adherence (IMA) — The IMA intervention is a shared-decision making intervention that promotes health literacy and patient participation in the decision making process during the recommendation and prescription of a new drug for the management of a cardiovascular disease and diabetes.
  The IMA intervention has four main components: training for healthcare professionals (general practitioners (GP), nurses and community pharmacists) on non-initiation, shared-decision making, health literacy and use of decision aids; intervention decision aids (leaflets and website); implementation of the IMA intervention during the GP's consultation; and information support provided by the nurses and community pharmacists that will use the intervention decision aids to explore the patients's doubts and harmonise and standardise the discourse between primary healthcare professionals.
  Arms: Initial Medication Adherence (IMA) intervention
Other: Usual care — Health professionals in the usual care group will prescribe medication and provide information as usual.
  Arms: Usual care

SUMMARY:
The purpose of this study is to assess the effectiveness and the cost-effectiveness of the Initial Medication Adherence (IMA) Intervention.

DETAILED DESCRIPTION:
A pragmatic cluster randomised control trial will be conducted to evaluate the effectiveness of the IMA intervention in comparison to usual care, in the increase of initiation of medicines for CVD and diabetes (antihypertensive, lipid-lowering, antidiabetic and antiplatelet medications) prescribed in Primary Care (PC). The impact of the IMA intervention on secondary adherence and clinical indicators will be evaluated.

A multicenter pragmatic RCT, with cluster allocation and 2 parallel branches (IMA intervention vs. usual care) based on health records or RWD will be conducted.

PC centres' personnel, including general practitioners (GP), nurses and community pharmacists, from different areas around Catalonia (Spain), will be cluster randomised 1:1 into intervention and control groups, stratified according to the type of PC centre, either rural or urban and taking into consideration the size and localization of the PC centre and the main predictors of non-initiation (socioeconomic status, mean age, % immigrant population of the PC centre).

The IMA intervention will provide clinicians with knowledge, skills and tools to help the patient make an informed decision. PC centre personnel in the intervention group will receive training on medication non-initiation, communication abilities, health literacy, shared decision making and the use of support tools such as leaflets and the IMA website.

ELIGIBILITY:
Inclusion Criteria:

* Primary Care health professionals and pharmacists who:
* Agree to participate in the clinical trial and process evaluation.
* Attend the training course
* Are not plannig to be on sick leave during the study period (e.g. maternity leave).
* Patients who:
* Are prescribed a new treatment of cardiovascular disease o diabetes by a doctor who participates in the clinical trial.
* Are >18 years old
* Do not reject to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4153 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Initiation | 1 month and 3 months after recruitment
  Patients who receive a new prescription (a prescription is considered new if there is no previouos prescription from the same group in the previous 6 months) will be considered initiators if they fill-up their prescription in the community pharmacy.
  Prescription and dispensation databases will be compared to classify prescriptions as initiated and non-initiated.

SECONDARY OUTCOMES:
Rate of adherence | 1 year after recruitment
  Adherence will be calculated based on the Medication Possesion Ratio (MPR is the sum of the days' supply for all fills of a given drug in a particular time period, divided by the number of days in the time period).
Reduction of Cardiovascular Risk | 1 year after recruitment
  Framingham risk score will be calculated.

OTHER OUTCOMES:
Visits to primary care | 1 year after recruitment
  Number of visits to primary care will be counted from electronic health records.
Visits to secondary care | 1 year after recruitment
  Number of visits to secondary care will be counted from electronic health records.
Visits to emergency room | 1 year after recruitment
  Number of visits to ER will be counted from electronic health records.
Use of diagnostic tests | 1 year after recruitment
  Number of diagnostic tests used will be counted from electronic health records.
Hospital admissions | 1 year after recruitment
  Number of inpatient and outpatient hospital admissions will be counted from electronic health records.
Use of medication | 1 year after recruitment
  Number of medication boxes dispensed will be counted from electronic health records.
Productivity loss | 1 year after recruitment
  Sick leaves used as a proxy for productivity loss, counted from electronic health records.
Cardiovascular events | 1 year after recruitment
  All incident events during follow-up, classified according to the International Classification of Diseases, 10th version (ICD10) collected in electronic health records. The events of interest include: Diabetes (E10-E14); dislipidemia (E78); hypertensive diseases (I10-I15); Ischemic heart diseases (I20-I25); other heart diseases (I50, I51); cerebrovascular diseases (I60-I69); diseases of arteries (I70-I79); glomerular diseases (N03, N08) and Acute kidney failure and chronic kidney disease (N17-N19).
Rate of Mortality | 1 year after recruitment
  mortality data from electronic health records

CONTACTS AND LOCATIONS:
Locations (24):
- Spain (24):
  - CAP Pou Torre, Begues, Barcelona
  - CAP Calaf, Calaf, Barcelona
  - CAP Corbera de Llobregat, Corbera de Llobregat, Barcelona
  - CAP La Llagosta, La Llagosta, Barcelona
  - CAP Martorell, Martorell, Barcelona
  - CAP Montornès del Vallès, Montornès del Vallès, Barcelona
  - CAP Ripollet, Ripollet, Barcelona
  - CAP Vinyets, Sant Boi de Llobregat, Barcelona
  - Parc Sanitari Sant Joan de Déu, Sant Boi de Llobregat, Barcelona
  - CAP Sant Sadurni d'Anoia, Sant Sadurní d'Anoia, Barcelona
  - CAP Sant Vicenç de Castellet, Sant Vicenç de Castellet, Barcelona
  - CAP Sitges, Sitges, Barcelona
  - CAP Montcada i Reixac, Montcada i Reixac, Barcelon
  - CAP Sort, Sort, Lleida
  - CAP de Tremp, Tremp, Lleida
  - CAP Cornudella de Montsant, Cornudella de Montsant, Tarragona
  - CAP Sant Pere, Reus, Tarragona
  - CAP Santa Coloma de Queralt, Santa Coloma de Queralt, Tarragona
  - CAP Drassanes, Barcelona
  - CAP Horta, Barcelona
  - CAP La Marina, Barcelona
  - CAP Montilivi, Girona
  - CAP Sant Pere i Sant Pau, Tarragona
  - CAP Bonavista, Tarragona

IPD SHARING:
Plan to Share IPD: No
The research team is not the data owner as they are only re-using information that is the property of the public health institutions. Consequently, meta-data cannot be published by the authors nor data can be identified with a DOI.

REFERENCES:
- [Derived] Corral-Partearroyo C, Sanchez-Vinas A, Aznar-Lou I, Penarrubia-Maria MT, Gil-Girbau M, Gallardo-Gonzalez C, Olmos-Palenzuela MDC, Rubio-Valera M. Effectiveness of a patient-centred complex intervention to improve Initial Medication Adherence to cardiovascular disease and diabetes treatments in primary care (the IMA-cRCT study): a pragmatic cluster randomised controlled trial using real-world data. BMJ Qual Saf. 2025 Jul 1:bmjqs-2024-018402. doi: 10.1136/bmjqs-2024-018402. Online ahead of print. PMID 40592577
- [Derived] Corral-Partearroyo C, Sanchez-Vinas A, Penarrubia-Maria MT, Gil-Girbau M, Aznar-Lou I, Palma-Vasquez C, Gallardo-Gonzalez C, Olmos-Palenzuela MDC, Rubio-Valera M. Implementation of a patient-centred complex intervention to improve Initial Medication Adherence to cardiovascular disease and diabetes treatments in primary care (the IMA-cRCT study): a mixed-methods process evaluation. BMJ Qual Saf. 2025 Jun 8:bmjqs-2024-018403. doi: 10.1136/bmjqs-2024-018403. Online ahead of print. PMID 40484629
- [Derived] Corral-Partearroyo C, Sanchez-Vinas A, Gil-Girbau M, Penarrubia-Maria MT, Aznar-Lou I, Gallardo-Gonzalez C, Olmos-Palenzuela MDC, Rubio-Valera M. Complex multidisciplinary intervention to improve Initial Medication Adherence to cardiovascular disease and diabetes treatments in primary care (the IMA-cRCT study): mixed-methods process evaluation protocol. BMJ Open. 2022 Oct 31;12(10):e067468. doi: 10.1136/bmjopen-2022-067468. PMID 36316078
- [Derived] Sanchez-Vinas A, Corral-Partearroyo C, Gil-Girbau M, Penarrubia-Maria MT, Gallardo-Gonzalez C, Olmos-Palenzuela MD, Aznar-Lou I, Serrano-Blanco A, Rubio-Valera M. Effectiveness and cost-effectiveness of an intervention to improve Initial Medication Adherence to treatments for cardiovascular diseases and diabetes in primary care: study protocol for a pragmatic cluster randomised controlled trial and economic model (the IMA-cRCT study). BMC Prim Care. 2022 Jul 5;23(1):170. doi: 10.1186/s12875-022-01727-6. PMID 35790915